CLINICAL TRIAL: NCT03956654
Title: A Phase IV Study to Collect Data on the Efficacy and Safety of RIBociclib With Letrozole in Older Women (≥70 Years) With HR+ and HER2- Advanced Breast Cancer (aBC) With no Prior Systemic Therapy for Advanced Disease.
Brief Title: A Phase IV Study to Collect Data on the Efficacy and Safety of RIBociclib in Older Women With Breastcancer
Acronym: RibOB
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Hans Wildiers, adjunct head of clinic, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s61033
Record Dates: First submitted 2019-04-12; First posted 2019-05-21 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; elderly; geriatric assessment; geriatric oncology; translational research; biomarkers
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected at T0 (i.e. at the time of inclusion of the patient), at T1 (i.e. at day 15 of the first treatment cycle) and at T2 (after 3 months) and in addition to routine laboratory exams, blood drawn will be processed and frozen for future translational research exploring biological aging markers (as predictive markers of functional decline and survival) and biomarkers of response prediction. The central biobanking laboratory in Leuven will provide complete blood sampling sets per patient, containing 3 subsets (one for each time point) with all blood tubes, pre-printed labels and serum/plasma aliquot vials required at that time point, as well as disposable Pasteur pipettes for serum/plasma transfer.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ribociclib — combination of ribociclib and letrozole
  Other Names: Kisqali

SUMMARY:
The RibOB study is a prospective, open lable, single arm trial which will evaluate the clinical efficacy, overall safety and tolerability of ribociclib in combination with letrozole in older women (≥70 years) with HR+/HER2- aBC and no prior hormonal treatment for advanced disease (as per approved indication).

DETAILED DESCRIPTION:
The RibOB study is an observational prospective, open lable single arm phase IV trial which will evaluate the clinical efficacy, overall safety and tolerability of ribociclib in combination with letrozole in older women (≥70 years) with HR+, HER2- advanced breast cancer and no prior hormonal treatment for advanced disease as per the indication approved by the European Medicines Authority (EMA) and as made available by Belgian national authorities in the national health care system. A total of maximum 150 patients will be enrolled for treatment with Letrozole (2.5 mg once daily) + ribociclib 600 mg (day 1 to 21 in a 28 day cycle), which will continue until disease progression, intolerable toxicity or patient/physician decision to withdraw. During the study, patients will be continuously evaluated for disease progression as per national standard of care (approximately every 12 weeks radiologically); for safety; and for quality of life and geriatric assessment components including functional status with QoL assessment and CGA at 3 months (+/- 2 weeks) and at 1 year (+/-2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patient is a female ≥ 70 years old at the time of informed consent.
* Advanced breast cancer (defined as locoregionally recurrent or metastatic not amenable to curative therapy).
* Histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by local laboratory (defined as ER and/or PgR ≥1% or Allred >2).
* HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test as determined by local laboratory testing according to ASCO-CAP guidelines is necessary.
* Patient has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by local laboratory), preferably tested a maximum of 14 days before enrolment:
* Patient has signed informed consent obtained before any trial-related activities and according to local guidelines.
* Subjects must be able to communicate with the investigator and comply with the requirements of the study procedures.

Exclusion Criteria:

* Patient has a known hypersensitivity to any of the excipients of ribociclib or letrozole.
* Patients who received any CDK4/6 inhibitor previously.
* Patient who received any prior systemic antihormonal therapy or chemotherapy for advanced breast cancer.
* Patient is concurrently using other systemic anti-cancer therapy (except bone modifying agents).
* Patient with central nervous system (CNS) metastases and/or documented meningeal carcinomatosis unless they meet ALL the following criteria:
* At least 4 weeks from prior therapy for CNS disease completion (including radiation and/or surgery) to starting the study treatment;
* Clinically stable CNS lesions at the time of study treatment initiation and not receiving steroids and/or enzyme-inducing anti-epileptic medications for the management of brain metastases for at least 2 weeks (radiological confirmation of brain disease status is not necessary).
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol: (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* Patients who already have or who are at significant risk of developing QTc prolongation are not eligible for the study. This includes patients:
* with long QT syndrome;
* with uncontrolled or significant cardiac disease, including recent myocardial infarction, congestive heart failure, unstable angina and bradyarrhythmias;
* with electrolyte abnormalities (potassium, magnesium, sodium and calcium) that are NCI CTCAE 4.03 grade 2 or higher (for details, see table 10 ). Note: phosphate testing is not mandatory, but should the investigator consider measuring it before enrolment, the same rules may be applied

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study will include older women (defined as ≥70 years) with HR+, HER2- advanced breast cancer who had not received any prior hormonal agent for treatment of advanced disease. It is expected that at least 50% of patients will be older than 75 years.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2018-2022
  Clinical efficacy: Progression-free survival (PFS) (defined as the length of time from the start of treatment and death or progression of disease) as determined by the local investigator using RECIST 1.1 rules.

SECONDARY OUTCOMES:
Time to treatment failure (TTF) | 2018-2022
  Efficacy: Time to treatment failure (TTF). It is defined as time from date of start of treatment to the date of event defined as the first documented progression, death due to any cause or withdrawal from treatment.
Overall response rate (ORR) | 2018-2022
  Efficacy: Overall response rate (ORR), for patients with measurable disease as determined locally by investigator according to RECIST 1.1. It is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.
Overall Survival (OS) | 2018-2022
  Efficacy: Overall survival (OS). It is defined as the length of time from the start of treatment and death from any cause.
Breast cancer specific survival (BCSS) | 2018-2022
  Efficacy: Breast cancer specific survival (BCSS). It is defined as the length of time from the start of treatment and death from breast cancer.
Adverse events | 2018-2022
  Safety: Incidence of Adverse Events according to the NCI-CTCAE 4.03 during study treatment and according to the results of baseline CGA evaluation; Number of patients who stop ribociclib before progression ; number of patients needing dose interruption/reduction.
Treatment discontinuation | 2018-2022
  Safety: Number of patients who stop ribociclib before progression
Treatment interruption | 2018-2022
  Safety: number of patients needing dose interruption
Treatment reduction | 2018-2022
  Safety: number of patients needing dose reduction
PFS / OS | 2018-2022
  Prediction Modeling I: PFS and OS prognostic model based on clinical/pathologic characteristics
CGA / QoL | 2018-2022
  Prediction Modeling II: Baseline CGA and QoL and relation with PFS/OS
Quality of Life (1) | 2018-2022
  Evolution of QoL during study treatment: EORTC QLQ-C30 (modified) and EORTC IL15 questionnaires
Quality of Life (2) | 2018-2022
  Correlation of baseline QoL with OS
Quality of Life (3) | 2018-2022
  Correlation of baseline QoL with toxicity grade III-IV
Comprehensive Geriatric Assessment | 2018-2022
  Evolution of CGA during study treatment
Plasma Biomarker Research (1) | 2018-2022
  Evolution of potential aging biomarkers during study treatment, and predictive value of baseline aging biomarkers on toxicity, PFS and OS (correcting for the prognostic metastatic index in PFS / OS)
Plasma Biomarker Research (2) | 2018-2022
  Predictive capacity of thymidine kinase on toxicity, PFS, OS and RR (correcting for the prognostic metastatic index in PFS, OS and RR). Thymidine kinase d1 versus d15 drop, and Thymidine kinase d15 level
Plasma Biomarker Research (3) | 2018-2022
  Develop a plasma microRNA signature for response to study treatment (pre-dose cycle 3)
Plasma Biomarker Research (4) | 2018-2022
  Evaluation of plasma antitumor immunity induction by study treatment at day 15 of cycle 1.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Wildiers, prof. dr., Study Chair — UZ Gasthuisberg
Locations (1):
- UZ Gasthuisberg Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided